CLINICAL TRIAL: NCT07286253
Title: A Single-arm, Multicenter Phase II Clinical Study of QL1706 Plus Chemotherapy as Neoadjuvant Therapy for Locally Advanced Cervical Cance
Brief Title: QL1706 Plus Chemotherapy as Neoadjuvant Therapy for Locally Advanced Cervical Cancer: A Phase II Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Lipai Chen, Chief physician, Affiliated Cancer Hospital & Institute of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL-CC-QIBA-3005
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Neoadjuvant Treatment for Locally Advanced Cervical Cancer
MeSH Terms: interventions — Infusions, Intravenous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: QL1706 plus nab-paclitaxel plus cisplatin/carboplatin (Experimental)
  Interventions: Drug: Drug: Drug: QL1706 5mg/kg, iv drip,d1,Q3W;Albumin-Bound Paclitaxel 260mg/m2, iv drip, d1, Q3W;Cisplatin50mg/m2, iv drip, d1, Q3W;Carboplatin AUC 5 ivdrip, d1, Q3W

INTERVENTIONS:
Drug: Drug: Drug: QL1706 5mg/kg, iv drip,d1,Q3W;Albumin-Bound Paclitaxel 260mg/m2, iv drip, d1, Q3W;Cisplatin50mg/m2, iv drip, d1, Q3W;Carboplatin AUC 5 ivdrip, d1, Q3W — Drug: Drug: QL1706 5mg/kg, iv drip,d1,Q3W;Albumin-Bound Paclitaxel 260mg/m2, iv drip, d1, Q3W;Cisplatin50mg/m2, iv drip, d1, Q3W;Carboplatin AUC 5 ivdrip, d1, Q3W

SUMMARY:
Cervical cancer ranks as the second most common malignancy of the female genital tract. According to the World Health Organization, there are 530,000 new cases and approximately 250,000 cervical-cancer-related deaths worldwide each year, with 80% of these deaths occurring in women from developing countries. Early-stage disease can be managed surgically, whereas advanced or recurrent cervical cancer is treated with individualized multimodal therapy; nevertheless, the optimal management of locally advanced cervical cancer (FIGO 2018 stage IB3-IIA2) remains controversial. Chemoradiation is standard, but neoadjuvant chemotherapy followed by radical surgery after tumor down-staging is also used. More than 90% of cervical cancers are driven by persistent infection with high-risk human papillomavirus (HPV), which evades host immunity in part by up-regulating PD-L1 on tumor cells. Published series report PD-L1 positivity in 34.4-96% of cervical cancers, with even higher rates in squamous-cell histology, providing a rationale for PD-1/PD-L1 blockade. QL1706, a novel bispecific immunotherapeutic agent, has recently been approved as monotherapy for second-line treatment of advanced cervical cancer.QL1706, developed by Qilu Pharmaceutical using the proprietary MabPair™ platform, is the first bispecific antibody simultaneously targeting PD-1 and CTLA-4, showing synergistic anti-tumor activity and favorable tolerability.Unlike previous phase II/III trials of PD-1 monotherapy, this study does not restrict enrolment to patients with PD-L1-positive tumors, so QL1706 is expected to confer benefit in the second-line management of recurrent or metastatic cervical cancer. Therefore, investigating QL1706-based combination regimens as neoadjuvant treatment for treatment-naïve disease is also highly relevant and may improve outcomes in women with locally advanced cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* (1) Has given written informed consent (or consent provided by an immediate family member if the subject is unable to do so) after full explanation of the study.

  (2) Female, aged ≥ 18 and ≤ 70 years on the date of informed-consent signature. (3) Histologically confirmed cervical cancer: A. Squamous-cell carcinoma, adenocarcinoma, or adenosquamous carcinoma; B. Previously untreated-no prior anti-cancer therapy for cervical cancer; C. FIGO 2018 stage IB3 or IIA2; D. Stage IIICr without involvement of the lower third of the vagina and without parametrial infiltration.

  (4) At least one measurable lesion by CT or MRI per RECIST 1.1. Note: Lesions situated in a prior radiation field or previously treated by local-regional therapy must be classified as non-target lesions unless clear progression is documented or tumor viability is confirmed by biopsy, and no other measurable lesion exists; in that case the lesion may serve as a target lesion.

  (5) Archival tumor tissue obtained within 5 years before enrollment OR a freshly obtained biopsy (≈ 7 unstained FFPE slides, minimum 5; preference for recent sample).

The biopsied lesion must not be selected as a RECIST 1.1 target lesion unless no other site is suitable and the biopsy was performed outside the screening period. If a subject cannot provide the required slides and the investigator judges re-biopsy to be unsafe, the number of slides may be reduced at the investigator's discretion.

(6) Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1. (7) Life expectancy ≥ 12 weeks. (8) Adequate function of major organs documented within 14 days before randomisation (no transfusion, albumin, recombinant human thrombopoietin or colony-stimulating factors allowed during this period): Haematology Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L Platelets ≥100 × 10⁹/L Haemoglobin ≥90 g/L Hepatic Total bilirubin ≤1.5 × upper limit of normal (ULN) ALT and AST ≤2.5 × ULN (≤5 × ULN if liver metastases present) Serum albumin ≥30 g/L Renal Serum creatinine ≤1.5 × ULN; OR if >1.5 × ULN, calculated creatinine clearance ≥60 mL/min (Cockcroft-Gault) Coagulation APTT ≤1.5 × ULN PT/INR ≤1.5 × ULN Cardiac Left-ventricular ejection fraction (LVEF) ≥50% Urinalysis Dipstick proteinuria <2+ If ≥2+, 24-hour urine protein must be <1.0 g to permit entry (9) Women of child-bearing potential must use a highly effective contraceptive method from informed-consent signature until 180 days after the last study-dose administration and must not be pregnant or lactating.

Exclusion Criteria:

* (1) Prior exposure to any immunotherapy, including immune-checkpoint inhibitory antibodies (e.g., anti-PD-1, anti-PD-L1, anti-CTLA-4), immune-checkpoint agonistic antibodies (e.g., anti-ICOS, CD40, CD137, GITR, OX40), or cellular immunotherapy.

  (2) Systemic or severe infection requiring intravenous antibiotics for >7 days within 2 weeks before enrolment, or unexplained fever >38.5 °C detected during screening or within 2 weeks prior to enrolment (fever judged by the investigator to be tumour-related is permitted).

  (3) Systemic corticosteroids (>10 mg/day prednisone or equivalent) or other immunosuppressive agents (e.g., cyclophosphamide, azathioprine, methotrexate, thalidomide, TNF-α inhibitors) for any indication within 2 weeks before enrolment. Topical, nasal or inhaled corticosteroids are allowed; systemic steroids given solely for prophylaxis of contrast allergy are also permitted.

  (4) Treatment with immunomodulatory agents such as thymosin, lentinan, interferon or interleukins within 2 weeks before enrolment.

  (5) Use within 2 weeks before enrolment of aspirin (>325 mg/day), clopidogrel (>75 mg/day), dipyridamole, ticlopidine, cilostazol, or any therapeutic-dose anticoagulant other than low-molecular-weight heparin.

  (6) Use of modern Chinese herbal preparations approved by NMPA for anti-cancer therapy within 2 weeks before enrolment.

  (7) Major surgery, open biopsy or significant traumatic injury within 4 weeks before enrolment; or planned elective major surgery during the study. Local invasive procedures (e.g., core biopsy) within 1 week before enrolment are excluded, except for vascular-access device placement.

  (8) Anti-cancer therapy (chemotherapy, endocrine therapy, targeted therapy, biological therapy, trans-arterial chemo-embolisation, etc.) within 4 weeks before enrolment.

  (9) Symptomatic CNS metastases, leptomeningeal disease or spinal-cord compression at baseline. Asymptomatic subjects with stable CNS disease who have completed any prior CNS-directed therapy ≥2 weeks earlier and have been off corticosteroids and anti-convulsants for ≥2 weeks may be enrolled.

  (10) Clinically significant hydronephrosis that cannot be relieved by nephrostomy or ureteral stenting.

  (11) Recurrent third-space fluid (e.g., pleural effusion or ascites) requiring repeated drainage and judged poorly controlled.

  (12) Active or potentially relapsing autoimmune disease, except: vitiligo, alopecia, psoriasis or eczema not requiring systemic therapy; hypothyroidism due to autoimmune thyroiditis on stable hormone replacement; or type 1 diabetes on stable-dose insulin.

  (13) History of gastrointestinal or genitourinary perforation/fistula, or intra-abdominal abscess within 6 months before enrolment (subjects are eligible if the underlying defect has been surgically corrected).

  (14) Bowel obstruction within 6 months before enrolment (subjects with incomplete obstruction that has resolved after treatment may be enrolled at the investigator's discretion), active intra-abdominal inflammation (including but not limited to peptic ulcer, diverticulitis or colitis).

  (15) Clinically significant cardiovascular disorders:
  1. Myocardial infarction, unstable angina, pulmonary embolism or other arterial/venous thrombo-embolic or cerebrovascular event requiring medical intervention within 6 months before enrolment;
  2. NYHA class III-IV congestive heart failure;
  3. Serious arrhythmia requiring medication;
  4. Mean QTcF >470 ms on 12-lead ECG (Fridericia formula) at screening. (16) Co-existing conditions that would increase the risk of adverse events during the study:

  <!-- -->

  1. Poorly controlled hypertension (systolic >150 mmHg and/or diastolic >100 mmHg) despite optimal therapy;
  2. Prior hypertensive crisis or hypertensive encephalopathy;
  3. History of intracranial or spinal haemorrhage;
  4. Bleeding diathesis, severe coagulopathy (off anticoagulation) or tumour encasing major vessels;
  5. Haemoptysis ≥½ teaspoon bright-red blood per episode, radiation enteritis/colitis or radiation cystitis with bleeding within 3 months before enrolment;
  6. Evidence of free intra-abdominal air;
  7. Serious non-healing or dehiscent wound or untreated fracture;
  8. Any other condition judged by the investigator to confer unacceptable risk. (17) Interstitial lung disease, pneumoconiosis, drug-related pneumonitis or severely impaired pulmonary function that might interfere with detection or management of suspected drug-related pulmonary toxicity.

     (18) HIV-positive; active hepatitis B (HBsAg-positive and HBV-DNA >500 IU/mL, or above local lower limit of detection if >500 IU/mL); active hepatitis C (subjects with positive HCV antibody but HCV-RNA below local lower limit of detection are eligible).

     (19) Known active tuberculosis; known active syphilis. (20) Other active malignancy within 5 years before informed consent, except adequately treated localised cancers (e.g., basal- or squamous-cell skin cancer, superficial bladder cancer, ductal carcinoma in situ of the breast).

     (21) Prior allogeneic haematopoietic stem-cell or organ transplantation (corneal transplant allowed).

     (22) Live-vaccine administration within 4 weeks before enrolment. (23) Participation in another clinical trial and receipt of an investigational product within 4 weeks before enrolment.

     (24) History of substance abuse (drugs or alcohol) or psychiatric/neurological disorder (epilepsy, dementia, hepatic encephalopathy, etc.) that could compromise compliance.

     (25) Known hypersensitivity to macromolecular protein preparations, or contraindication/allergy to any component of QL1706, cisplatin/carboplatin or paclitaxel.

     (26) Any condition that, in the opinion of the investigator, could increase study-related risk or interfere with interpretation of results.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) | 2 years
  Pathological complete response (pCR) is defined as the absence of residual malignant tumor cells in the resected specimen.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 years
  The ratio of patients who are evaluated as CR or PR
Disease-free survival (DFS) | 2 years
  defined as the time from enrollment to the first documented disease progression or death from any cause, whichever occurs first.
2-year disease-free survival rate (2-year DFS rate) | 2 years
  2-year disease-free survival rate (2-year DFS rate): defined as the proportion of participants who remain alive and without radiologically documented disease progression at 2 years from enrollment.

CONTACTS AND LOCATIONS:
Locations (1):
- Lipai Chen, Guangzhou, Guangdong, China